CLINICAL TRIAL: NCT04783883
Title: Electrical Vestibular Nerve Stimulation (VeNS): A Follow-up Safety Assessment of Long-Term Usage
Brief Title: Electrical Vestibular Nerve Stimulation (VeNS): A Follow-up Assessment of Long-term Usage
Status: Completed | Type: Observational
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: R D Gardi Medical College, Ujjain (Unknown)
Responsible Party: Sponsor
Other Study IDs: RWDMES01
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Safety Issues
Keywords: Neuromodulation; Safety; Vestibular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vestal DM — Battery powered non-invasive neurostimulation device (1.5mA)

SUMMARY:
A follow-up assessment study of the long-term safety of vestibular electrical stimulation as delivered by the Vestal DM Device.

DETAILED DESCRIPTION:
A retrospective, open-label, follow-up study assessing the long-term safety and efficacy of vestibular electrical stimulation as delivered by the Vestal DM Device.

ELIGIBILITY:
Inclusion Criteria:

* Vestal DM user (more than 6 months)

Exclusion Criteria:

* Vestal DM device user (less than 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vestal DM device users from any country.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Assessment of hearing function as reported by formal audiometry testing | Baseline
  Formal audiometry testing to be conducted using the AMTAS Flex Device

SECONDARY OUTCOMES:
Frequency of device related adverse events | Baseline
Inspection of the skin behind the ears (mastoid area) | Baseline
  Photographic inspection of the skin behind the ears to confirm no skin irritation has been caused at the mastoid area where the electrode pads are placed
Otoscope examination of the inside of both ear canals and tympanic membranes | Baseline
  Photographs to be taken of both ear canals and both tympanic membranes using the Awelor Wireless Smart Otoscope (Model Number: T1).

CONTACTS AND LOCATIONS:
Locations (1):
- Neurovalens Ltd., 7 James St. South, Belfast, United Kingdom